CLINICAL TRIAL: NCT04788667
Title: Effectiveness of a Health Education Programme as a Preventive Treatment for Chronic Migraine: A Randomized Clinical Trial
Brief Title: Effectiveness of a Health Education Programme for Prevention of Chronic Migraine: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Universidad San Jorge (Other); Hospital Clínico Universitario Lozano Blesa (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, PT, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Migraine2021
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chronic Migraine
Keywords: chronic migraine; Telerehabilitation; Prophylaxis; Exercise Therapy; Education
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A health education programme using a telerehabilitation platform
  Interventions: Other: A health education programme using a telerehabilitation platform
- Control Group (Active Comparator): General recommendations using a telerehabilitation platform
  Interventions: Other: A health education programme using a telerehabilitation platform

INTERVENTIONS:
Other: A health education programme using a telerehabilitation platform — All patients enrolled in the study will receive information through the tele rehabilitation platform, although the experimental group will have specific training/education whereas the control group will only receive some general recommendations as control/sham
  Other Names: Regular pharmacological treatment provided by their neurologists (Fremanezumab o Erenumab); Regular pharmacological treatment provided by their neurologists (Botulinum Toxin)

SUMMARY:
Chronic migraine (CM) is a common and frequent disorder, which has a major impact on the quality of life of migraine sufferers, interfering with physical function, productivity at work, personal life and leisure, lifestyle and psychological well-being.

The use of a prophylactic drug treatment is recommended if headache is present more than 8 days per month. In addition, several studies have shown benefits of non-pharmacological interventions such as self-management strategies, manual therapy and exercise. However, no studies have been found that analyse the beneficial effect of a combination of a preventive drug treatment and a health education programme.

Thus, this project would offer a service of health education through a telerehabilitation programme for patients with chronic migraine under prophylactic drug treatment.

The aim of this study is to compare the combination of a prophylactic drug therapy and a health education programme in the preventive treatment of patients with chronic migraine.based on the hypothesis that a health education program for chronic migraine patients could decrease the number of migraine days.

DETAILED DESCRIPTION:
Design:

A randomised, double-blind, controlled clinical trial will be conducted in two parallel groups, in which all patients with migraine chronic are receiving prophylactic drug treatment with Fremanezumab or Erenumab as prescribed by a physician. Moreover, patients in the experimental group will receive a health education programme and patients in the control group will receive a programme of general recommendations.

Intervention:

A 4-week baseline data collection period is included to record the frequency and intensity of migraine pain before starting the study.

The intervention will be carried out for 6 months with a follow-up at 1, 3 and 12 months.

Experimental group:

Patients will receive health education through video-tutorials that can be watched on the HEFORA platform. Each video-tutorial will contain the content of an educational session, including health information in the areas of pain education, migraine neurophysiology, relaxation techniques, sleep habits, eating habits, physical exercise, coping strategies and emotion management.

Control group:

Patients will receive video-tutorials with general recommendations though HEFORA platform.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-65 years.
* Patients diagnosed with CM following the ICHD-III criteria.
* Patients with migraine onset before the age of 50 years.
* Patients who have been diagnosed with chronic migraine for at least 1 year.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Women with menstrual migraine.
* Patients with severe or unstable psychiatric pathology that contraindicates the use of drug treatment.
* Allergic patients or those who show sensitivity to components of the drug treatment.
* Patients who refuse to sign the informed consent form or to participate in the study.
* Patients who decide not to continue in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Headache frequency (days/month) | baseline (30 days after intervention), month 1, month 2, month 3, month 4, month 5, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Changes in number of days/month of headache following the criteria of "The International Classification of Headache Disorders (ICHD-III). Headache frequency will be assessed with a headache diary.

SECONDARY OUTCOMES:
Headache intensity | baseline (30 days after intervention), month 1, month 2, month 3, month 4, month 5, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Changes in intensity of headache: 0, (no pain), 1 (mild), 2 (moderate) and 3 (intense).
  Both the maximum pain and the average pain for the month will be measured.
Analgesic medication | baseline (30 days after intervention), month 1, month 2, month 3, month 4, month 5, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Analgesic medication use (days/month).
The six-item Headache Impact Test (HIT-6) | pre-intervention (day 1), month 1, month 2, month 3, month 4, month 5, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Changes in the impact of headache. The HIT-6 measures the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning and psychological distress. The HIT-6 also measures the severity of headache pain. Each item is answered on a 5-point Likert scale (6 = never, 8 = rarely, 10 = sometimes, 11 = very often, 13 = always). The final score is obtained from simple summation of the six items.
Migraine Disability Assessment (MIDAS) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 9 (follow-up 2), month 12 (follow-up 3).
  Changes in headache-related disability. MIDAS questionnaire is a brief, self-administered questionnaire designed to quantify headache-related disability over a 3 month period. Once scored, the test gives the patient an idea of how debilitating his/her migraines are based on this scale: 0 to 5, MIDAS Grade I, Little or no disability; 6 to 10, MIDAS Grade II, Mild disability; 11 to 20, MIDAS Grade III, Moderate disability; 21+, MIDAS Grade IV, Severe disability.
Allodynia Symptom Checklist (ASC-12) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Changes in allodynia. ASC-12 assess frequency of cutaneous allodynia symptoms during headache attack, including 12 questions.
Pressure pain threshold (PPT) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Changes in PPT using an algometer (Wagner, FDX). To determine PPT, pressure was increased at a rate of approximately 1 kg/s and subjects were asked to say 'pain' at the point the sensation first became painful, at which point pressure was released and the readout recorded. Thresholds were taken as the average of two measures taken 30 s apart.
  * 21 scalp points used in the international standard of encephalography:
    o Fp2, Fp4, F8, C4, T4, P4, T6, C2, Fp1, F3, F7, C3, T3, P3, T5 y O1, Fpz, Fz, Cz, Pz y Oz.
  * Upper trapezius, bilaterally (midpoint between the C7 spine and the acromion).
  * Suboccipital area, bilaterally (the insertion of the suboccipital and upper trapezius muscle).
  * Control point, bilaterally (distally located in the muscle belly of the medial gastrocnemius).
Temporal summation (TS) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Changes in TS using Pin-Prick. The temporal summation assessment will be performed using a 256 mN "Pin-Prick" by performing 10 consecutive pressures of one second each with a pause interval of one second. The patient will then evaluate the intensity of pain on a visual analogue scale. It will be applied on a single point of the upper trapezius muscle.
Hospital Anxiety and Depression (HADS) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 12 (follow-up 3).
  Changes in depression and anxiety. The questionnaire comprises seven questions for anxiety and seven questions for depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Pain Catastrophizing Scale (PCS) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 12 (follow-up 3).
  Changes in catastrophism. The PCS is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). The PCS is broken into three subscales being magnification, rumination, and helplessness.
Tampa Scale for Kinesiophobia (TSK) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 12 (follow-up 3).
  Changes in kinesiophobia. TSK abbreviated version is 11 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance, scoring range from 1 (strongly disagree) to 4 (strongly agree).
International physical activity questionnaire (IPAQ) short-form. | pre-intervention (day 1), month 3, month 6 (post-intervention), month 12 (follow-up 3).
  Changes in physical activity. The IPAQ short-form consists of 8 items to estimate the time spent performing physical activities (moderate to vigorous) and inactivity (time spent sitting).
Pittsburg Sleep Quality Index (PSQI) | pre-intervention (day 1), month 3, month 6 (post-intervention), month 12 (follow-up 3).
  Changes in sleep quality. The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points.
Chronic Pain Self-efficacy Scale | pre-intervention (day 1), month 3, month 6 (post-intervention), month 12 (follow-up 3).
  Changes in self-efficacy. The 19-item Chronic Pain Self-efficacy Scale (CPSS) measures three domains of pain self-efficacy: pain management, physical functioning, and coping with symptoms. It consists of a Likert-type scale ranging from 0 (=I see myself as totally incapable) to 10 (=I see myself as totally capable).
Satisfaction scale | month 6 (post-intervention).
  Changes in satisfaction. A 5-point Likert-type scale will be used (1= Very dissatisfied; 2= Somewhat dissatisfied; 3=Indifferent; 4= Somewhat satisfied; 5= Very satisfied).
Pollutants | baseline (30 days after intervention), before intervention, month 1, month 2, month 3, month 4, month 5, month 6 (post-intervention), month 7 (follow-up 1), month 9 (follow-up 2), month 12 (follow-up 3).
  Pollutants measured through a wearable. It will measure different pollutants such as particulate matter (PM), ozone (O3), nitrogen dioxide (NO2) and sulphur dioxide (SO2).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Spain